CLINICAL TRIAL: NCT05658081
Title: Stapled Antimesenteric Functional End-to-end Anastomosis (Kono-S) Versus Stapled Antimesenteric Isoperistaltic Side-to-side Anastomosis for the Postoperative Recurrence of Crohn's Disease: a Randomized Control Trial Study
Brief Title: Comparison of Two Stapled Antimesenteric Anastomosis for CD: a Randomized Control Trial Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Zhu Weiming, Jinling Hospital, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: jinlingH20221202
Record Dates: First submitted 2022-12-02; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Crohn Disease; Recurrence
MeSH Terms: conditions — Crohn Disease; Recurrence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kono-S group (Experimental): patients in this arm will receive stapled Kono-S anastomosis after bowel resection
  Interventions: Procedure: Kono-S group
- Side-to-side group (Other): patients in this arm will receive stapled antimesenteric isoperistaltic side-to-side anastomosis after bowel resection
  Interventions: Procedure: Side-to-side group

INTERVENTIONS:
Procedure: Kono-S group — patients in this arm will receive stapled Kono-S anastomosis after bowel resection
  Arms: Kono-S group
Procedure: Side-to-side group — patients in this arm will receive stapled antimesenteric isoperistaltic side-to-side anastomosis after bowel resection
  Arms: Side-to-side group

SUMMARY:
The postoperative recurrence of Crohn's diseases (CD) remains high. Stapled anti-mesenteric functional end-to-end anastomosis was safe for CD patients. Its impact on the postoperative recurrence of CD was unknown. Whether it is superior than the conventional anastomosis (stapled antimesenteric isoperistaltic side-to-side anastomosis) needs explored. The trial aims to compare the different impacts of the two antimesenteric anastomosis configurations on the anastomotic recurrence following bowel resection.

ELIGIBILITY:
Inclusion Criteria:

* patients with Crohn's disease needing bowel resection and anastomosis;
* ileocolic anastomosis；
* written consent acquired

Exclusion Criteria:

* patients underwent enterostomy;
* small bowel anastomosis;
* anticipating other trial.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 236 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
the endoscopic recurrence rate at 1 year after surgery | at 1 year after surgery(6-18month)
  the endoscopic recurrence rate at 1 year after surgery

SECONDARY OUTCOMES:
the clinical recurrence rate at 1 and 5 year after surgery | 1 and 5 year after surgery
  the clinical recurrence rate at 1 and 5 year after surgery
the surgical recurrence rate at 1 and 5 year after surgery | 1 and 5 year after surgery
  the surgical recurrence rate at 1 and 5 year after surgery
the endoscopic recurrence rate at 1 year after surgery | 1 and 5 year after surgery
  the endoscopic recurrence rate at 1 year after surgery
quality of life for CD patients inflammatory bowel disease questionnaire(IBDQ) | 1 and 5 year after surgery
  IBDQ ， higher means better，IBDQ，7-224；
quality of life for CD patients Short Form 12 | 1 and 5 year after surgery
  Short Form 12 ， higher means better，Short Form-12， 0-12；

CONTACTS AND LOCATIONS:
Overall Officials: Yi Li, Ph.D, Principal Investigator — Jinling Hospital，Nanjing， China
Locations (1):
- Department of General Surgery, Jinling hosptal,Medical School of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No